CLINICAL TRIAL: NCT02249078
Title: A Multicenter, Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Sequential-Cohort, Multiple-Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of 3 Subcutaneous and 1 Intravenous Dose of E6011 in Subjects With Active Crohn's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of 3 Subcutaneous and 1 Intravenous Dose of E6011 in Subjects With Active Crohn's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6011-A001-102
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 100 mg subcutaneous once every 2 weeks with initial double dose (200 mg total)
  Interventions: Drug: E6011
- Cohort 2 (Experimental): 200 mg subcutaneous once every 2 weeks with initial double dose (400 mg total)
  Interventions: Drug: E6011
- Cohort 3 (Experimental): 400 mg subcutaneous once every 2 weeks with initial double dose (800 mg total)
  Interventions: Drug: E6011
- Cohort 4 (Experimental): 10 mg/kg IV at Day 1, Day 8, Day 15, and every 2 weeks thereafter
  Interventions: Drug: E6011
- Placebo (Placebo Comparator): Placebo 2-mL vial solution for injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6011 — E6011 solution for injection
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: Placebo — Placebo 2-mL vial solution for injection
  Arms: Placebo

SUMMARY:
This is a multicenter, Phase 1b, randomized, double-blind, placebo-controlled, sequential-cohort, multiple ascending dose (MAD) study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of 3 subcutaneous and 1 intravenous dose of E6011 in subjects with active Crohn's disease (CD). Thirty-two subjects will be randomized to one of 4 dose cohorts (8 per cohort) and will receive E6011 or placebo for 10 weeks. The first 3 cohorts will receive E6011 or placebo via subcutaneous injection and the last cohort will receive E6011 or placebo by intravenous injection. The ratio of E6011 to placebo within each cohort will be 3:1. The study has 2 phases: Prerandomization and Randomization.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Male or female subjects age greater than or equal to 18 years old at the time of informed consent
2. Confirmed diagnosis of CD, with at least one documented lesion within the reach of a colonoscope (terminal ileal or ileo-colonic or colonic) from a previous colonoscopy, for a minimum duration of 6 months at the time of screening
3. Active CD with a CD activity index (CDAI) score greater than or equal to 220 and less than or equal to 450
4. Colonoscopic evidence of CD involvement with active inflammation of terminal ileum and/or colon at Screening (performed only in subjects who have otherwise met all of the inclusion and none of the exclusion criteria)
5. Inadequate response to, loss of response to, or intolerance of at least one of the following agents as defined below:

   * Immunomodulators:
   * Signs and symptoms of persistently active disease despite a history of at least one 8-week regimen of oral azathioprine (AZA) (greater than or equal to 1.5 mg/kg) or 6-mercaptopurine (6-MP) mg/kg (greater than or equal to 0.75 mg/kg) OR
   * Signs and symptoms of persistently active disease despite a history of at least one 8-week regimen of methotrexate (MTX) (greater than or equal to 12.5 mg/week)
   * History of intolerance to at least 1 immunomodulator (including, but not limited to) nausea/vomiting, abdominal pain, pancreatitis, liver function test (LFT) abnormalities, lymphopenia, thiopurine methyltransferase (TPMT) genetic mutation, infection
   * Tumor Necrosis Factor (TNF)-alpha antagonists:
   * Signs and symptoms of persistently active disease despite a history of at least one 4-week induction regimen of one of the following agents:
   * Infliximab: 5 mg/kg IV, 2 doses at least 2 weeks apart
   * Adalimumab: one 80 mg SC dose followed by one 40-mg dose at least 2 weeks apart
   * Certolizumab pegol: 400 mg SC dose, 2 doses at least 2 weeks apart OR
   * Recurrence of symptoms during scheduled maintenance dosing following prior clinical benefit (discontinuation despite clinical benefit does not qualify)
   * History of intolerance to at least 1 TNF antagonist (including, but not limited to infusion-related reaction, demyelination, congestive heart failure, infection)
6. C-reactive protein greater than or equal to 5 mg/L at screening or fecal calprotectin greater than or equal to 250 ug/g
7. Females must not be breastfeeding or pregnant at Screening (as documented by a negative beta-human chorionic gonadotropin [B-hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
8. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 70 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 70 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 70 days after study drug discontinuation. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
9. Provide written informed consent
10. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal [other than CD], renal disease, active infection, vasculitides) that in the opinion of the investigator(s) could affect the patient's safety or interfere with the study assessments
2. Any neurologic abnormality at screening
3. A prolonged QT/QTc interval (QTc greater than 450 ms) as demonstrated by a repeated ECG at Screening
4. History of any severe allergy
5. Scheduled for surgery during planned participation in the study
6. Previous ileo-colonic resections or presence of an ostomy
7. Presence of active fistulizing CD
8. Total parenteral nutrition (TPN) or enema for treating CD within 2 weeks before Screening
9. Treatment with adalimumab or certolizumab within 2 weeks before Screening
10. Treatment with infliximab within 4 weeks (or 8 weeks if subjects received 10 mg/kg) before Screening
11. Treatment with vedolizumab (in case of approval or off-label use) or any other monoclonal antibody within 8 weeks before starting the study treatment
12. History of treatment with natalizumab
13. Changes in dose of 5-aminosalicylic acid, 6-MP, MTX, and AZA therapy within 4 weeks of Screening
14. Doses of greater than 30 mg/day of prednisone or equivalent at Screening
15. Parenteral corticosteroids use within 4 weeks of Screening
16. Treatment with cyclosporine (oral or IV), tacrolimus hydrate (excluding eyedrops or skin cream), sirolimus, or mycophenolate mofetil within 8 weeks before Screening
17. Positive Clostridium difficile toxin test at Screening
18. Known to be human immunodeficiency virus (HIV) positive at Screening
19. History of tuberculosis or known current active tuberculosis
20. Positive results for Mycobacterium tuberculosis using an Interferon-Gamma Release Assay at Screening
21. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
22. Use of live vaccine and immunoglobulin preparations within 12 weeks of screening
23. Cluster of differentiation-4 (CD4) positive cell count below 200/microliter (uL) or white blood cell count below 3,000/uL at screening
24. Any of the following laboratory abnormalities in tests conducted during Screening

    * Hemoglobin: less than 8.0 g/dL
    * Neutrophil count: less than 1,500/uL
    * Platelet count: less than 100,000/uL
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT): greater than 2.5 times the upper limit of standard reference values
    * Serum creatinine: greater than 1.5 mg/dL
25. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years
26. History of drug or alcohol dependency or abuse within the 2 years prior to Screening
27. Current use of illegal recreational drugs
28. Currently enrolled in another clinical study or used any investigational drug or device within 28 days preceding informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) as a measure of the short-term safety and tolerability of E6011 | Up to 3 years
  The short-term safety and tolerability of subcutaneous (SC) and intravenous (IV) doses of E6011 compared to placebo in subjects with active CD. Safety assessments will consist of monitoring and recording all AEs and SAEs; regulatory monitoring of hematology, blood chemistry, and urine values; periodic measurement vital signs and ECGs; and performance of physical examinations.

SECONDARY OUTCOMES:
Concentration of E6011 measured over time in blood samples. | Up to 3 years
The number and percentage of participants with anti-E6011 antibodies detected in blood samples over time. | Up to 3 years
The number of screen positives, confirm positives, and relative anti-E6011 levels measured in blood samples from participants. | Up to 3 years
Change from baseline in the percentage of immunohistochemical staining for the CX3CR1+ protein in intestinal tissue over time. | Up to 3 years